CLINICAL TRIAL: NCT02372357
Title: A New Dosing Regimen for Posaconazole Prophylaxis in Children Based in Body Surface Area
Brief Title: A New Dosing Regimen for Posaconazole Prophylaxis in Children Based on Body Surface Area
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Ap.r Kim Vanstraelen, PharmD, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2841/20 Feb 2012
Record Dates: First submitted 2015-02-06; First posted 2015-02-26 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Hematological Malignancy
Keywords: chemotherapy; stem cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posaconazole 120mg/m² tid (Experimental): Pediatric patients admitted to receive chemotherapy or hematopoietic stem cell transplantation for the treatment of a hematological malignancy are receiving Posaconazole prophylaxis 120 mg/m² tid.
  At steady state, blood sampling will be performed: 9 blood samples will be taken during 1 dosing interval to evaluate the pharmacokinetics of posaconazole.
  Interventions: Drug: Posaconazole prophylaxis 120 mg/m² tid; Procedure: Blood sampling

INTERVENTIONS:
Drug: Posaconazole prophylaxis 120 mg/m² tid — Patients are receiving posaconazole to prevent invasive fungal infections in a dose of 120 mg/m² tid
Procedure: Blood sampling — During steady state treatment with posaconazole (at least 7 days), 9 blood samples are taken via a central venous catheter to evaluate the pharmacokinetics of posaconazole.

SUMMARY:
A new prophylactic posaconazole dosing regimen of 120mg/m² tid is evaluated pharmacologically in children 13 years and younger, suffering from a hematologic malignancy.

DETAILED DESCRIPTION:
Invasive fungal infections (IFI), especially candidiasis and aspergillosis, are a serious threat to immunocompromised pediatric patients. Because diagnosis of IFI in pediatric patients is difficult, due to the lack of specific clinical and radiological signs and the low sensitivity of blood cultures, antifungal prophylaxis would largely optimize management of IFI in this setting. However, antifungal prophylaxis remains a matter of debate, as no clear consensus has yet been reached about the optimal drug. Very limited pediatric data are available, and current guidelines are mainly based on extrapolation of adult data. Fluconazole remains the drug of choice in many centers, despite its non-mould active spectrum. Itraconazole, liposomal amphotericin B and nebulized lipid-formulations of amphotericin B are often used off-label, although neither their pharmacokinetics (PK), nor their efficacy and safety have been documented in a proper way. Voriconazole is registered for children older than 2 years of age, mainly in the treatment setting. Moreover, its extremely variable PK profile, uncertainty about adequate exposure and risk for hepatotoxicity and neurotoxicity do not favor the use of voriconazole in this setting. Finally, micafungin only has low recommendation in the prophylactic setting, due to the possible risk of liver tumours.

Posaconazole would be the ideal antifungal drug to be used prophylactically in children for many reasons. It has a broad spectrum of activity, including emerging moulds like Aspergillus spp. and Zygomycetes. It has shown to be superior over fluconazole and itraconazole in preventing IFI in adults and it has a favorable safety profile, with nausea and vomiting being the most frequently encountered adverse events. However, lack of pharmacokinetic (PK) data in children younger than 13 years of age, results in only a marginal recommendation in current guidelines [8]. Little information is available about the correct dosing regimen of the available oral suspension in young pediatric patients, and similar to what is observed in adults, often very low posaconazole plasma concentrations (PPCs) are being measured. Therefore, therapeutic drug monitoring (TDM) is recommended to reach adequate PPCs above 0.5mg/L or 0.7 mg/L followed by increasing the dose as needed.

In this study, the pharmacokinetics of a newly introduced dosing regimen for posaconazole oral suspension is investigated, based on body surface area (BSA), used prophylactically in immunocompromised children under the age of 13.

Pediatric patients, admitted to the hospital to receive chemotherapy or hematopoietic stem cell transplantation are treated prophylactically with posaconazole 120mg/m² tid.

At steady state (after at least 7 days of posaconazole treatment), 9 plasma samples are collected in these patients to calculate the area under the curve and other relevant PK parameters as maximum and minimal plasma concentrations, volume of distribution, halflife and clearance rate.

Finally, these results will be compared to adult data in literature to evaluate whether 120mg/m² tid an adequate dosing regimen in children.

ELIGIBILITY:
Inclusion Criteria:

* 2-13 years of age
* hematological malignancy
* need for antifungal prophylaxis because of neutropenia caused by chemotherapy and/or hematopoietic stem cell transplantation.

Exclusion Criteria:

* <2 years of age
* > 13 years of age

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters of posaconazole | One day at steady state posaconazole treatment
  9 blood samples are taken during one day at steady state posaconazole plasma concentrations. The following pharmacokinetic parameters will be calculated using non-compartmental pharmacokinetic analysis: Cmax, Cmin, Tmax, Area Under the Curve during 1 dosing interval and over 24 hours, Clearance, Distribution volume, Halflife.

SECONDARY OUTCOMES:
Safety of posaconazole, focussing on nausea, vomiting and liver function abnormalities (according to the Common Terminology Criteria for Adverse Events (CTCAE classification). | patients will be followed for the duration of hospital stay, an expected average of 3-4 weeks
  Patients receiving posaconazole prophylactically are closely monitored for adverse events possibly related to the drug. They are clinically monitored for nausea, vomiting and diarrhea. Liver function abnormalities are scored according to the CTCAE classification.
Efficacy: patients are monitored for breakthrough infections according the the European Organisation for Research and Treatment of Cancer- Mycoses Study Group (EORTC-MSG) criteria. | patients will be followed for the duration of hospital stay, an expected average of 3-4 weeks
  Patients receiving posaconazole prophylactically are closely monitored for the presence of an invasive fungal infection. Patients are closely followed in case an invasive fungal infection is suspected: Fever is monitored, radiography is performed and galactomannan is measured frequently. Invasive fungal infections are categorized according to the revised EORTC-MSG criteria

CONTACTS AND LOCATIONS:
Overall Officials: Anca Colita, MD, Principal Investigator — Institutul Clinic Fundeni, Bucarest, Romania; Kim Vanstraelen, PharmD, Principal Investigator — Catholic University Leuven, Leuven, Belgium
Locations (2):
- Catholic University Leuven - Department of Pharmaceutical and Pharmacological Sciences, Leuven, Vlaams-Brabant, Belgium
- Institutul Clinic Fundeni, Bucharest, Sector 2, Romania